CLINICAL TRIAL: NCT03762005
Title: Peripheral Perfusion Versus Lactate Targeted Fluid Resuscitation in Septic Shock: ANDROMEDA-SHOCK PHYSIOLOGY STUDY
Brief Title: Peripheral Perfusion Versus Lactate Targeted Fluid Resuscitation in Septic Shock
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Comisión Nacional de Investigación Científica y Tecnológica (Other Government)
Responsible Party: Principal Investigator, Glenn Hernández, Titular Professor, Pontificia Universidad Catolica de Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 170323007
Record Dates: First submitted 2018-11-26; First posted 2018-12-03 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Septic Shock; Hyperlactatemia; Peripheral Perfusion
Keywords: Septic Shock; Lactate; Capillary refill time; Fluid Responsiveness; Mortality
MeSH Terms: conditions — Shock, Septic; Hyperlactatemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRT guided resuscitation (Experimental): Fluid resuscitation will be aimed at normalizing capillary refill time (CRT) during the intervention period. Fluid challenges will be administered at a rate of 500 ml of crystalloids over 30 minutes, with reassessment of CRT until achieving normal values, or the patient becomes fluid unresponsive, or a safety issue develops.
  Interventions: Other: CRT guided resuscitation
- Lactate guided resuscitation (Active Comparator): Fluid resuscitation will be aimed at normalizing or decreasing lactate levels by more than 20% every 2 hours during the intervention during the intervention period. Fluid challenges will be administered at a rate of 500 ml of crystalloids over 30 minutes, with reassessment of lactate every 2 hours until reaching target, or the patient becomes fluid unresponsive, or a safety issue develops.
  Interventions: Other: Lactate guided resuscitation

INTERVENTIONS:
Other: CRT guided resuscitation — Sequential approach with fluids (guided by dynamic predictors of fluid responsiveness), according to capillary refill time (CRT)
  Arms: CRT guided resuscitation
Other: Lactate guided resuscitation — Sequential approach with fluids (guided by dynamic predictors of fluid responsiveness), according to lactate levels
  Arms: Lactate guided resuscitation

SUMMARY:
Persistent hyperlactatemia has been traditionally considered as representing tissue hypoxia, and lactate normalization is recommended as a resuscitation target by the Surviving Sepsis Campaign (SSC). However, other sources contribute to hyperlactatemia such as sustained adrenergic activity and impaired lactate clearance. Only hypoperfusion-related hyperlactatemia might be reversed by optimizing systemic blood flow.

Fluid resuscitation (FR) is used to improve cardiac output (CO) in septic shock to correct hypoperfusion. Nevertheless, if persistent hyperlactatemia is not hypoxia-related, excessive FR could lead to flow overload. In addition, kinetics of recovery of lactate is relatively slow, and thus it might be a suboptimal target for FR.

Peripheral perfusion appears as a promising alternative target. Abnormal capillary refill time (CRT) is frequently used as trigger for FR in septic shock. Studies demonstrated the strong prognostic value of persistent abnormal peripheral perfusion, and some recent data suggest that targeting FR on CRT normalization could be associated with less fluid loading and organ dysfunctions. The excellent prognosis associated with CRT recovery, the rapid-response time to fluid loading, its simplicity, and its availability in resource-limited settings, constitute a strong background to promote studies evaluating its usefulness to guide FR .

The study hypothesis is that a CRT-targeted FR is associated with less positive fluid balances, organ dysfunctions, and at least similar improvement of tissue hypoperfusion or hypoxia, when compared to a lactate-targeted FR. To test this hypothesis, the investigators designed a clinical physiological, randomized controlled trial in septic shock patients. Recruited patients will be randomized to FR aimed at normalizing CRT or normalizing or decreasing lactate >20% every 2 h during the study period. Fluid challenges (500 ml in 30 min intervals) will be repeated until perfusion target is achieved, or dynamic predictors of fluid responsiveness become negative, or a safety limit is reached. The design of our study is aimed at: a) determining if CRT targeted resuscitation is associated with less fluid resuscitation and fluid balances; b) determining if this strategy is associated with less organ dysfunctions; and c) if it results in similar improvement in markers of tissue hypoperfusion or hypoxia such as hepato-splanchnic blood flow or microcirculatory perfusion.

DETAILED DESCRIPTION:
GENERAL OBJECTIVE To demonstrate that a CRT-targeted FR is associated with less positive fluid balances, organ dysfunctions, and similar improvement of markers of tissue hypoperfusion and hypoxia, when compared to a lactate- targeted FR.

SPECIFIC OBJECTIVES

1. To determine if normalization of CRT is associated with less fluid resuscitation and positive 24-h fluid balances as compared to lactate-targeted resuscitation.
2. To determine if normalization of CRT is associated with less organ dysfunctions as compared to lactate-targeted resuscitation.
3. To determine if CRT-targeted resuscitation compared to lactate-targeted resuscitation leads to similar improvement in markers of tissue hypoperfusion or hypoxia at the end of fluid resuscitation
4. To determine if normality of all the selected hypoperfusion variables (central venous oxygen saturation (ScvO2), central venous to arterial carbon dioxide pressure difference (P(cv-a)CO2), and CRT) at different time-points in septic shock patients can predict the absence of tissue hypoperfusion and hypoxia.

For this Research Project, several variables of tissue hypoperfusion that can only be assessed by special perfusion-monitoring techniques were included.

Sublingual microcirculatory assessment: Sublingual microcirculatory alterations have been well described in septic shock patients. Functional capillary density and microvascular blood flow are decreased, while heterogeneity is markedly enhanced. These alterations have been shown to be prognostic, with a rapid improvement in survivors but a progressive decline in nonsurvivors. A microcirculatory flow index (MFI) ≤ 2.5 and a proportion of perfused vessels (PPV) < 80% will be considered as categorical of microcirculatory hypoperfusion Liver blood flow: Plasma disappearance rate (PDR) of indocyanine green (ICG), with a non-invasive transcutaneous assessment of ICG clearance. Normal range is 18% to 25% per minute with a value < 15%/min categorically abnormal.

Muscle tissue O2 saturation: Muscle tissue O2 saturation (StO2). A decrease in this variable to <70% suggests profound tissue hypoperfusion.

Assessment of tissue hypoxia: There are two clinically calculable variables that have been proposed as closely representing tissue hypoxia: the venous- arterial CO2 (Cv- aCO2) to arterial-venous O2 content (Da-vO2) difference ratio (Cv- aCO2/Da-vO2) and the lactate/pyruvate (L/P) ratio . Both ratios are an expression of anaerobic metabolism at the cellular level and thus can be linked to hypoxia. For this research project, these variables were considered to ascertain the presence and resolution of tissue hypoxia.

* Cv-aCO2/Da-vO2 ratio: This ratio might be useful as a surrogate of the respiratory quotient. A ratio ≥ 1.4 could identify anaerobic CO2 generation. A high Cv-aCO2/Da-vO2 ratio in the setting of hyperlactatemia may favor anaerobic metabolism as the possible source of lactate, while a normal Cv-aCO2/Da-vO2 ratio suggesting that lactate accumulation is due to non-hypoperfusion- related causes.
* L/P ratio: In anaerobic conditions, pyruvate is transformed to lactate and thus the L/P ratio increases to ≥ 18. The L/P ratio is considered to be one of the most reliable indexes of hypoxia in critically ill patients.

METHODOLOGY A randomized controlled study of parallel groups was designed: Group A with a CRT-targeted fluid resuscitation strategy and group B with a lactate-targeted one.

This prospective study will be performed at the Hospital of the Pontifical Catholic University and at the Public Hospital of the South of Santiago, Chile.

The study was approved by the Institutional Review Board of both centers. A signed informed consent will be asked to the next of kin of all eligible patients, and confirmed by the patients when feasible.

The study intervention period will be of 6 hours I. Randomization A randomization sequence with an allocation of 1:1 will be generated by a computer program. Study-group assignment will be performed by means of randomized permuted blocks of eight. Allocation concealment will be maintained by means of central randomization.

Fluid challenges (500 ml of Ringer's lactate administered in 30 min intervals) are repeated until the perfusion target is normalized, or fluid responsiveness becomes negative, or a safety limit of an increase in central venous pressure (CVP) ≥ 5 mmHg after a fluid bolus is reached. The perfusion target in group A is a normal CRT ≤3 sec. The perfusion target in group B is an arterial lactate ≤ 2 mmol/l or a decrease >20% every 2h.

CRT will be assessed every 30 minutes and lactate every 2 hours during the 6h study intervention period, after which the treatment is liberalized for attending physicians.

If fluid resuscitation is stopped because the perfusion target is normalized, the time is registered, and the patient subjected to the specific research-related assessment protocol and followed until hospital discharge.

II. General management algorithm Besides sepsis source aggressive management, all patients will be treated according to our local algorithm aimed at macrohemodynamic stabilization and improvement of hypoperfusion. The algorithm has been described elsewhere. Co-interventions will be registered and considered in statistical analysis.

III. Specific research-related assessments For the purposes of this research protocol, several variables will be periodically measured or calculated as follows: at baseline, at 2h, at 6h and at 24h.

1. Macrohemodynamic variables such as mean arterial pressure,M, heart rate, norepinephrine dose, CVP, dynamic predictors.
2. Continuous cardiac output (CO) monitoring: this will be performed with non-invasive pulse-contour CO assessment acquired with this project (PiCCO device).
3. Metabolic-perfusion variables such as arterial lactate, ScvO2, and P(cva)CO2.
4. Peripheral perfusion assessment: CRT and mottling score
5. Sublingual microcirculation: It will be assessed with the side dark field (SDF) device. At each assessment, at least five 10-20 sec video images will be recorded. The analysis will be performed by eye following recent recommendations . From image analysis the following variables will be calculated (i) proportion of perfused vessels; (ii) microcirculatory flow index (MFI); All these indexes will be calculated separately for small (<20 microm diameter) and large vessels (> 20 microm diameter) .
6. Liver blood flow: An ICG finger clip well be fixed in every patient and then connected to a liver function monitor (LiMON; Pulsion Medical Systems, Munich, Germany). A dose of 0.25 mg/kg of ICG (LiMon Pulsion Medical Systems, Germany) will be injected through a central venous catheter.
7. Near infrared spectroscopy (NIRS): StO2 will be measured by a tissue spectrometer (InSpectra Model 325; Hutchinson Tc, Mn, USA). A NIRS probe will be placed on the skin of the thenar eminence
8. Ccv-aCO2/Da-vO2 ratio: This ratio will be calculated after taking arterial and central venous blood gases with the Douglas formula.
9. L/P ratio: This ratio will be assessed at 0, 6 and 24h during the study period, at baseline and when fluid resuscitation is stopped. Arterial blood samples for pyruvate will be taken and processed in our laboratory before 3h according to the method described by De Backer et al , including immediate deproteinization of the sample and analysis by enzymatic fluorometric-assay (Sigma-Aldrich, USA)
10. Sequential organ failure assessment (SOFA) at baseline, 24, 48 and at 72h . Finally, all patients will be followed until hospital discharge, and all data including demographic aspects, sepsis sources and management, inflammatory biomarkers, and severity scores and major outcomes will be registered.

STATISTICAL ANALYSIS Sample size calculation: the simple size calculation was based in some small clinical studies. In a recent study, a resuscitation strategy guided by peripheral perfusion offered important benefits in terms of fluid administration at 6 hours (4227 ± 1081 ml vs 6069 ± 1715 ml) and organ dysfunction, when compared with standard fluid therapy. In consequence, a 1600 ml difference in the mean 24-h total fluid administration between the experimental CRT group and the conventional lactate group was considered to be the critical threshold for hypothesis testing. If there is truly no difference between the standard and experimental treatment, then 46 patients are required (23 patients per arm) to be 90% sure that the lower limit of a two-sided confidence interval will be above the limit of -1600 mL at an alpha level of 0.05. Statistical analysis Intention to treat analysis will be performed in order to minimize bias.

Analyses will be performed as follows: Specific Objective #1: between study groups, the amount of fluids administered at the end of fluid resuscitation, and at 6, 24, 48 and 72h will be compared exclusively at each time-point with t-test, and comprehensively using ANOVA. Total 24-h fluid balance will be compared using t-test. Specific Objective #2, the status of peripheral perfusion normalization will be assessed in a categorical way (normal/abnormal) with chi-square at specific time-points (at the end of fluid resuscitation, 6, and 24h), and with means of SOFA score at each time-point up to 72h using t-test or Wilcoxon rank sum test if appropriate. A total comparison using ANOVA will be also performed. In the same line, the relative change of SOFA among time-points (with baseline value as the reference) and between study groups will be assessed with analysis of proportions, using the binomial distribution. Specific Objective #3: comparison of improvement on markers of tissue hypoperfusion and hypoxia between study groups will be mainly assessed in a categorical way using chi-square at different time-points, since those markers are qualitatively attributed a dichotomic normal/abnormal status. For some of them (ICG, StO2) as continuous variables, t-test or Wilcoxon rank sum test will be used at specific time points (at the end of fluid resuscitation, 6, 24h), and ANOVA for a global analysis. Specific Objective #4: For this objective, pooled data from all the studied patients will be used. Pearson correlations between selected hypoperfusion variables (ScvO2, P(cv-a)CO2, and CRT) with markers of tissue hypoperfusion/hypoxia will be explored at different time-points.

All statistical calculations will be performed using Stata Statistical Software, Release 14 (College Station, TX). A probability value (p-value) of less than 0.05 will be considered

ELIGIBILITY:
Inclusion Criteria:

* Septic shock diagnosed at ICU admission according to the Sepsis-3 Consensus Conference [35], basically septic patients with hypotension requiring norepinephrine (NE) to maintain a mean arterial pressure (MAP) of 65 mmHg, and serum lactate levels > 2 mmol/l after initial fluid resuscitation.
* Less than 24 h after fulfilling criteria for septic shock
* Positive fluid responsiveness assessment

Exclusion Criteria:

* 1. Pregnancy
* Anticipated surgery or dialytic procedure during the first 6h after septic shock diagnosis
* Do-not-resuscitate status
* Child B or C liver cirrhosis
* Active bleeding
* Severe concomitant acute respiratory distress syndrome (ARDS)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Amount of resuscitation fluids | at six hours
  The total amount of fluids administered as fluid challenges from baseline to 6 hours after starting protocol

SECONDARY OUTCOMES:
Total fluid balance | at 24 hours
  Balance of fluids in the first 24h (inputs-outputs)
Multiple organ dysfunction | At 24 hours, 48 hours and 72 hours
  Sequential Organ Failure Assessment (SOFA) scores assessed at baseline, 24 hours, 48 hours and 72 hours. The scale range is from 0 points to 24 points, where 0 points represent normality and no organ dysfunction, and 24 points severe organ dysfunction for the six organs evaluated. More than 10 points is considered severe organ dysfunction.
  The six organs evaluated in the Sequential Organ Failure Assessment score are: lungs, cardiovascular system, coagulation, liver, kidneys, and central nervous system. All six organs are evaluated from 0 (normal function) to 4 (severe dysfunction) and these sub-scores are summed to get the total SOFA score.
Sublingual microcirculation | at baseline, 6 hours and 24 hours
  Evaluation of sublingual microcirculation by SDF: Videos will be taken at the sublingual mucosa with the SDF device. Two parameters will be calculated systematically by off-line video analysis according to consensus recommendations: MFI (normal value 3.0, with <2.5 considered as abnormal (range 0-3); and PPV where 100% is normal, with <80% representing clear abnormalities (range 0-100%)
Hepato-splanchnic blood flow | At baseline, 6 hours and 24 hours
  Evaluation of hepato-splanchnic blood flow by ICG clearance: calculation of plasma dissapearance of ICG with normal values >18% in 15 minutes
Muscle tissue oxygenation | At baseline, 6 hours and 24 hours
  Evaluation of muscle tissue oxygen saturation by NIRS (normal value >75%)
Ccv-aCO2/Da-vO2 ratio | At baseline, 6 hours and 24 hours
  Assessed by the Ccv-aCO2/Da-vO2 ratio as a marker of tissue hypoxia: normal value <1
Lactate/Pyruvate ratio | At baseline, 6 hours and 24 hours
  Assessed by the L/P ratio as another marker of tissue hypoxia. Normal value 10

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Hernandez, PhD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Pontificia Universidad Catolica de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Vincent JL, De Backer D. Circulatory shock. N Engl J Med. 2014 Feb 6;370(6):583. doi: 10.1056/NEJMc1314999. No abstract available. PMID 24499231
- [Result] Cecconi M, De Backer D, Antonelli M, Beale R, Bakker J, Hofer C, Jaeschke R, Mebazaa A, Pinsky MR, Teboul JL, Vincent JL, Rhodes A. Consensus on circulatory shock and hemodynamic monitoring. Task force of the European Society of Intensive Care Medicine. Intensive Care Med. 2014 Dec;40(12):1795-815. doi: 10.1007/s00134-014-3525-z. Epub 2014 Nov 13. PMID 25392034
- [Result] Dougnac AL, Mercado MF, Cornejo RR, Cariaga MV, Hernandez GP, Andresen MH, Bugedo GT, Castillo LF; Grupo Chileno del Estudio de la Sepsis. [Prevalence of severe sepsis in intensive care units. A national multicentric study]. Rev Med Chil. 2007 May;135(5):620-30. doi: 10.4067/s0034-98872007000500010. Epub 2007 Jul 9. Spanish. PMID 17657331
- [Result] Hernandez G, Bruhn A, Castro R, Regueira T. The holistic view on perfusion monitoring in septic shock. Curr Opin Crit Care. 2012 Jun;18(3):280-6. doi: 10.1097/MCC.0b013e3283532c08. PMID 22473257
- [Result] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb S, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including The Pediatric Subgroup. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock, 2012. Intensive Care Med. 2013 Feb;39(2):165-228. doi: 10.1007/s00134-012-2769-8. Epub 2013 Jan 30. PMID 23361625
- [Result] Garcia-Alvarez M, Marik P, Bellomo R. Sepsis-associated hyperlactatemia. Crit Care. 2014 Sep 9;18(5):503. doi: 10.1186/s13054-014-0503-3. PMID 25394679
- [Result] Tapia P, Soto D, Bruhn A, Alegria L, Jarufe N, Luengo C, Kattan E, Regueira T, Meissner A, Menchaca R, Vives MI, Echeverria N, Ospina-Tascon G, Bakker J, Hernandez G. Impairment of exogenous lactate clearance in experimental hyperdynamic septic shock is not related to total liver hypoperfusion. Crit Care. 2015 Apr 22;19(1):188. doi: 10.1186/s13054-015-0928-3. PMID 25898244
- [Result] Hernandez G, Pedreros C, Veas E, Bruhn A, Romero C, Rovegno M, Neira R, Bravo S, Castro R, Kattan E, Ince C. Evolution of peripheral vs metabolic perfusion parameters during septic shock resuscitation. A clinical-physiologic study. J Crit Care. 2012 Jun;27(3):283-8. doi: 10.1016/j.jcrc.2011.05.024. Epub 2011 Jul 27. PMID 21798706
- [Result] Centers for Disease Control (CDC). Ectopic pregnancy--United States, 1987. MMWR Morb Mortal Wkly Rep. 1990 Jun 22;39(24):401-4. No abstract available. PMID 2112685
- [Result] Hernandez G, Bruhn A, Castro R, Pedreros C, Rovegno M, Kattan E, Veas E, Fuentealba A, Regueira T, Ruiz C, Ince C. Persistent Sepsis-Induced Hypotension without Hyperlactatemia: A Distinct Clinical and Physiological Profile within the Spectrum of Septic Shock. Crit Care Res Pract. 2012;2012:536852. doi: 10.1155/2012/536852. Epub 2012 Apr 18. PMID 22570774
- [Result] Hernandez G, Regueira T, Bruhn A, Castro R, Rovegno M, Fuentealba A, Veas E, Berrutti D, Florez J, Kattan E, Martin C, Ince C. Relationship of systemic, hepatosplanchnic, and microcirculatory perfusion parameters with 6-hour lactate clearance in hyperdynamic septic shock patients: an acute, clinical-physiological, pilot study. Ann Intensive Care. 2012 Oct 15;2(1):44. doi: 10.1186/2110-5820-2-44. PMID 23067578
- [Result] Hernandez G, Boerma EC, Dubin A, Bruhn A, Koopmans M, Edul VK, Ruiz C, Castro R, Pozo MO, Pedreros C, Veas E, Fuentealba A, Kattan E, Rovegno M, Ince C. Severe abnormalities in microvascular perfused vessel density are associated to organ dysfunctions and mortality and can be predicted by hyperlactatemia and norepinephrine requirements in septic shock patients. J Crit Care. 2013 Aug;28(4):538.e9-14. doi: 10.1016/j.jcrc.2012.11.022. Epub 2013 Apr 6. PMID 23566729
- [Result] Hernandez G, Bruhn A, Luengo C, Regueira T, Kattan E, Fuentealba A, Florez J, Castro R, Aquevedo A, Pairumani R, McNab P, Ince C. Effects of dobutamine on systemic, regional and microcirculatory perfusion parameters in septic shock: a randomized, placebo-controlled, double-blind, crossover study. Intensive Care Med. 2013 Aug;39(8):1435-43. doi: 10.1007/s00134-013-2982-0. Epub 2013 Jun 6. PMID 23740284
- [Result] Ospina-Tascon GA, Bautista-Rincon DF, Umana M, Tafur JD, Gutierrez A, Garcia AF, Bermudez W, Granados M, Arango-Davila C, Hernandez G. Persistently high venous-to-arterial carbon dioxide differences during early resuscitation are associated with poor outcomes in septic shock. Crit Care. 2013 Dec 13;17(6):R294. doi: 10.1186/cc13160. PMID 24330804
- [Result] Ospina-Tascon GA, Umana M, Bermudez W, Bautista-Rincon DF, Hernandez G, Bruhn A, Granados M, Salazar B, Arango-Davila C, De Backer D. Combination of arterial lactate levels and venous-arterial CO2 to arterial-venous O 2 content difference ratio as markers of resuscitation in patients with septic shock. Intensive Care Med. 2015 May;41(5):796-805. doi: 10.1007/s00134-015-3720-6. Epub 2015 Mar 20. PMID 25792204
- [Result] Ospina-Tascon GA, Umana M, Bermudez WF, Bautista-Rincon DF, Valencia JD, Madrinan HJ, Hernandez G, Bruhn A, Arango-Davila C, De Backer D. Can venous-to-arterial carbon dioxide differences reflect microcirculatory alterations in patients with septic shock? Intensive Care Med. 2016 Feb;42(2):211-21. doi: 10.1007/s00134-015-4133-2. Epub 2015 Nov 17. PMID 26578172
- [Result] Hernandez G, Tapia P, Alegria L, Soto D, Luengo C, Gomez J, Jarufe N, Achurra P, Rebolledo R, Bruhn A, Castro R, Kattan E, Ospina-Tascon G, Bakker J. Effects of dexmedetomidine and esmolol on systemic hemodynamics and exogenous lactate clearance in early experimental septic shock. Crit Care. 2016 Aug 2;20(1):234. doi: 10.1186/s13054-016-1419-x. PMID 27480413
- [Result] Malbrain ML, Marik PE, Witters I, Cordemans C, Kirkpatrick AW, Roberts DJ, Van Regenmortel N. Fluid overload, de-resuscitation, and outcomes in critically ill or injured patients: a systematic review with suggestions for clinical practice. Anaesthesiol Intensive Ther. 2014 Nov-Dec;46(5):361-80. doi: 10.5603/AIT.2014.0060. PMID 25432556
- [Result] Hernandez G, Luengo C, Bruhn A, Kattan E, Friedman G, Ospina-Tascon GA, Fuentealba A, Castro R, Regueira T, Romero C, Ince C, Bakker J. When to stop septic shock resuscitation: clues from a dynamic perfusion monitoring. Ann Intensive Care. 2014 Oct 11;4:30. doi: 10.1186/s13613-014-0030-z. eCollection 2014. PMID 25593746
- [Result] Marik PE. Iatrogenic salt water drowning and the hazards of a high central venous pressure. Ann Intensive Care. 2014 Jun 21;4:21. doi: 10.1186/s13613-014-0021-0. eCollection 2014. PMID 25110606
- [Result] Gu WJ, Zhang Z, Bakker J. Early lactate clearance-guided therapy in patients with sepsis: a meta-analysis with trial sequential analysis of randomized controlled trials. Intensive Care Med. 2015 Oct;41(10):1862-3. doi: 10.1007/s00134-015-3955-2. Epub 2015 Jul 8. No abstract available. PMID 26154408
- [Result] Jansen TC, van Bommel J, Schoonderbeek FJ, Sleeswijk Visser SJ, van der Klooster JM, Lima AP, Willemsen SP, Bakker J; LACTATE study group. Early lactate-guided therapy in intensive care unit patients: a multicenter, open-label, randomized controlled trial. Am J Respir Crit Care Med. 2010 Sep 15;182(6):752-61. doi: 10.1164/rccm.200912-1918OC. Epub 2010 May 12. PMID 20463176
- [Result] Jones AE, Shapiro NI, Trzeciak S, Arnold RC, Claremont HA, Kline JA; Emergency Medicine Shock Research Network (EMShockNet) Investigators. Lactate clearance vs central venous oxygen saturation as goals of early sepsis therapy: a randomized clinical trial. JAMA. 2010 Feb 24;303(8):739-46. doi: 10.1001/jama.2010.158. PMID 20179283
- [Result] Puskarich MA, Trzeciak S, Shapiro NI, Albers AB, Heffner AC, Kline JA, Jones AE. Whole blood lactate kinetics in patients undergoing quantitative resuscitation for severe sepsis and septic shock. Chest. 2013 Jun;143(6):1548-1553. doi: 10.1378/chest.12-0878. PMID 23740148
- [Result] Bakker J, de Backer D, Hernandez G. Lactate-guided resuscitation saves lives: we are not sure. Intensive Care Med. 2016 Mar;42(3):472-474. doi: 10.1007/s00134-016-4220-z. Epub 2016 Feb 1. No abstract available. PMID 26831675
- [Result] Vallee F, Vallet B, Mathe O, Parraguette J, Mari A, Silva S, Samii K, Fourcade O, Genestal M. Central venous-to-arterial carbon dioxide difference: an additional target for goal-directed therapy in septic shock? Intensive Care Med. 2008 Dec;34(12):2218-25. doi: 10.1007/s00134-008-1199-0. Epub 2008 Jul 8. PMID 18607565
- [Result] Lima A, Bakker J. Clinical assessment of peripheral circulation. Curr Opin Crit Care. 2015 Jun;21(3):226-31. doi: 10.1097/MCC.0000000000000194. PMID 25827585
- [Result] van Genderen ME, Engels N, van der Valk RJ, Lima A, Klijn E, Bakker J, van Bommel J. Early peripheral perfusion-guided fluid therapy in patients with septic shock. Am J Respir Crit Care Med. 2015 Feb 15;191(4):477-80. doi: 10.1164/rccm.201408-1575LE. No abstract available. PMID 25679107
- [Result] Hernandez G, Teboul JL. Is the macrocirculation really dissociated from the microcirculation in septic shock? Intensive Care Med. 2016 Oct;42(10):1621-1624. doi: 10.1007/s00134-016-4416-2. Epub 2016 Jun 11. No abstract available. PMID 27289357
- [Result] Brunauer A, Kokofer A, Bataar O, Gradwohl-Matis I, Dankl D, Bakker J, Dunser MW. Changes in peripheral perfusion relate to visceral organ perfusion in early septic shock: A pilot study. J Crit Care. 2016 Oct;35:105-9. doi: 10.1016/j.jcrc.2016.05.007. Epub 2016 May 12. PMID 27481743
- [Result] Hernandez G, Bruhn A, Ince C. Microcirculation in sepsis: new perspectives. Curr Vasc Pharmacol. 2013 Mar 1;11(2):161-9. PMID 23506495
- [Result] Vellinga NA, Boerma EC, Koopmans M, Donati A, Dubin A, Shapiro NI, Pearse RM, Machado FR, Fries M, Akarsu-Ayazoglu T, Pranskunas A, Hollenberg S, Balestra G, van Iterson M, van der Voort PH, Sadaka F, Minto G, Aypar U, Hurtado FJ, Martinelli G, Payen D, van Haren F, Holley A, Pattnaik R, Gomez H, Mehta RL, Rodriguez AH, Ruiz C, Canales HS, Duranteau J, Spronk PE, Jhanji S, Hubble S, Chierego M, Jung C, Martin D, Sorbara C, Tijssen JG, Bakker J, Ince C; microSOAP Study Group. International study on microcirculatory shock occurrence in acutely ill patients. Crit Care Med. 2015 Jan;43(1):48-56. doi: 10.1097/CCM.0000000000000553. PMID 25126880
- [Result] Ospina-Tascon GA, Hernandez G, Cecconi M. Understanding the venous-arterial CO2 to arterial-venous O2 content difference ratio. Intensive Care Med. 2016 Nov;42(11):1801-1804. doi: 10.1007/s00134-016-4233-7. Epub 2016 Feb 12. No abstract available. PMID 26873834
- [Result] Rimachi R, Bruzzi de Carvahlo F, Orellano-Jimenez C, Cotton F, Vincent JL, De Backer D. Lactate/pyruvate ratio as a marker of tissue hypoxia in circulatory and septic shock. Anaesth Intensive Care. 2012 May;40(3):427-32. doi: 10.1177/0310057X1204000307. PMID 22577907
- [Result] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Result] Monnet X, Teboul JL. Assessment of volume responsiveness during mechanical ventilation: recent advances. Crit Care. 2013 Mar 19;17(2):217. doi: 10.1186/cc12526. No abstract available. PMID 23510457
- [Result] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239
- [Result] Castro R, Regueira T, Aguirre ML, Llanos OP, Bruhn A, Bugedo G, Dougnac A, Castillo L, Andresen M, Hernandez G. An evidence-based resuscitation algorithm applied from the emergency room to the ICU improves survival of severe septic shock. Minerva Anestesiol. 2008 Jun;74(6):223-31. Epub 2008 Mar 21. PMID 18356807
- [Derived] Castro R, Kattan E, Ferri G, Pairumani R, Valenzuela ED, Alegria L, Oviedo V, Pavez N, Soto D, Vera M, Santis C, Astudillo B, Cid MA, Bravo S, Ospina-Tascon G, Bakker J, Hernandez G. Effects of capillary refill time-vs. lactate-targeted fluid resuscitation on regional, microcirculatory and hypoxia-related perfusion parameters in septic shock: a randomized controlled trial. Ann Intensive Care. 2020 Nov 2;10(1):150. doi: 10.1186/s13613-020-00767-4. PMID 33140173